CLINICAL TRIAL: NCT02333253
Title: Delayed Start vs Conventional Antagonist Protocol in Poor Responders Pretreated by Estradiol in Luteal Phase.
Brief Title: Delayed Start Versus Conventional Antagonist Protocol in Poor Responders Pretreated by Estradiol in Luteal Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Other Complications Associated With Artificial Fertilization
Keywords: poor responders; GnRH antagonist; Conventional protocol
MeSH Terms: interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delayed start protocol (Active Comparator): First group received 300 U r FSH +150 U urinary GN from day 2 till day of HCG ,dose adjusted according to the response then 0.25 cetrotide S.c was added on when leading follicle reach >12 mm, HCG was given only if we have at least 3 mature follicles >14 mm and the leading one >17mm then OPU done after 36 hrs of HCG, oocytes were denuded and fertilized by ICSI to avoid low fertilization rate by conventional IVF,embryo transfer were done on day 3 when we have at least one embryo GI other wise cancelled ET, then cyclogest 800mg were given intravaginal for 14 days then quantitative BHCG done and considered positive if > 5miu/ML
  Interventions: Drug: cetrotide
- conventional antagonist protocol (Active Comparator): Second group were received cetrotide 0.25 mg s.c alone from day 2 to day 8then we initiate GN therapy by same initial GN dose (300FSH+150U urinary GN).same adjustment of dose were done and antagonist restarted when DF >12mm, till day of HCG, OPU done after 36 hrs of HCG, oocytes were denuded and fertilized by ICSI to avoid low fertilization rate by conventional IVF,embryo transfer were done on day 3 when we have at least one embryo GI other wise cancelled ET, then cyclogest 800mg were given intravaginal for 14 days then quantitative BHCG done and considered positive if > 5miu/ML
  Interventions: Drug: cetrotide

INTERVENTIONS:
Drug: cetrotide — 0.25 cetrotide S.c was added on when leading follicle reach >12 mm
  Other Names: cetrorelix acetate

SUMMARY:
40 patients attending IVF center during 2013 &2014 were fulfilling criteria of poor response and they failed to go through OPU as they gave <3 mature follicles on a dose of 300U GN or more. All patients were revised for history, examinations and investigations, including age, type and duration of infertility, day 3 FSH, Day 3 E2, AMH, AFC.

DETAILED DESCRIPTION:
40 patients attending IVF center during 2013 &2014 were fulfilling criteria of poor response and they failed to go through OPU as they gave <3 mature follicles on a dose of 300U GN or more. All patients were revised for history, examinations and investigations, including age, type and duration of infertility, day 3 FSH, Day 3 E2, AMH, AFC All patients were 35 years old ore more We exclude patient >44ys ,AMH <0.3ng/ml,FSH >13, also patients of DM, endometriosis, general disease were excluded, any local uterine anomalies were excluded.

All patients received OCP for one cycle Then all had taken estradiol tablet 2 mg for one week prior to menses of the test cycle from Day 21 to day 28 Then we divide them into 2 groups US were done to exclude any cyst or follicle >10mm First group received 300 U r FSH +150 U urinary GN from day 2 till day of HCG,dose adjusted according to the response then 0.25 cetrotide S.c was added on when leading follicle reach >12 mm, HCG was given only if we have at least 3 mature follicles >14 mm and the leading one >17mm then OPU done after 36 hrs of HCG, oocytes were denuded and fertilized by ICSI to avoid low fertilization rate by conventional IVF,embryo transfer were done on day 3 when we have at least one embryo GI other wise cancelled ET, then cyclogest 800mg were given intravaginal for 14 days then quantitative BHCG done and considered positive if > 5miu/ML 28 day after ET, TVS was done to confirm ongoing pregnancy by visualization of IU sac.

Second group were received cetrotide 0.25 mg s.c alone from day 2 to day 8then we initiate GN therapy by same initial GN dose (300FSH+150U urinary GN).same adjustment of dose were done and antagonist restarted when DF >12mm, till day of HCG, HCG,OPU, ET were done by same method and under same criteria, luteal support and follow were the same.

ELIGIBILITY:
Inclusion Criteria:

1 Poor responders 2. Age >35 years

Exclusion Criteria:

1. patient >44ys ,
2. AMH <0.3ng/ml,
3. FSH >13, also
4. patients of DM ,endometriosis ,general disease were excluded,
5. any local uterine anomalies were excluded.

Ages: 35 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
oocyte retrieved number | Induction cycle an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt